CLINICAL TRIAL: NCT04863079
Title: Pembrolizumab for Adjuvant Treatment After R0 Resection of Thoracic ESCC Patients With Lymph Node Positive: A Single-arm, Open-label, PhaseⅡTrial
Brief Title: Pembrolizumab in Post Radical Operation ESCC Patients With Lymph Node Positive ( KEYSTONE-004 )
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20210220A
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: ESCC; Adjuvant Treatment; Lymph Node Positive; Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab for Postoperative Adjuvant Treatment of ESCC (Experimental): Participants receive pembrolizumab 200 mg IV, Q3W, up to one year or disease progression or intolerance as postoperative adjuvant treatment of ESCC with pN+.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Pembrolizumab 200 mg IV, Q3W, up to one year or disease progression or intolerance.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of postoperative adjuvant treatment of pembrolizumab in patients with thoracic esophageal squamous cell carcinoma （ESCC） who have not received neoadjuvant therapy before undergoing R0 resection, and have positive postoperative lymph nodes.

DETAILED DESCRIPTION:
For patients with thoracic esophageal squamous cell carcinoma （ESCC） who have undergone R0 resection, have not received neoadjuvant therapy, and have positive postoperative lymph nodes, there is no international consensus on whether postoperative adjuvant therapy is required. The JCOG9204 study reported that for patients with ESCC with positive lymph nodes after R0 resection, postoperative adjuvant chemotherapy can improve the disease-free survival (DFS) of the ESCC patients. However, due to the adverse effects of chemotherapy, patients are often difficult to tolerate. We designed a single-arm, open-label, phase II trial of pembrolizumab for adjuvant treatment after R0 resection of thoracic ESCC Patients with lymph node positive. The purpose of this study is to observe and evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ESCC;
2. Patients have not received neoadjuvant therapy.
3. Thoracic ESCC with R0 resection and positive postoperative lymph nodes;
4. Have a performance status of 0 or 1 on the ECOG Performance Scale;
5. Age 18-70 years old, both men and women;
6. Be willing and able to provide written informed consent/assent for the trial;
7. Demonstrate adequate organ function , all screening labs should be performed within 10 days of treatment initiation;
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
9. Be willing to provide postoperative tissue specimens. After tumor recurrence, continue to be willing to provide tissue samples such as needle biopsy.

Exclusion Criteria:

1. Neoadjuvant therapy (radiotherapy, immunotherapy, or chemotherapy) for ESCC;
2. Non-R0 resection for ESCC;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs);
5. Has severe hypersensitivity and adverse events (≥Grade 3) to pembrolizumab and/or any PD-1/PD-L1 inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  Time from the enrollment to death of any cause
Disease-free survival (DFS) | 24 months
  Time from the enrollment to disease relapse after complete resection or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, MD, PhD, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No